CLINICAL TRIAL: NCT00924768
Title: A Study of Inhalation of 20,000 EU CCRE and MCC in Otherwise Healthy Individuals Who Are Current Cigarette Smokers
Brief Title: A Study of Inhalation of 20,000 EU CCRE and Mucociliary Clearance (MCC) in Otherwise Healthy Individuals Who Are Current Cigarette Smokers
Acronym: IRB 09-0259
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, David B. Peden, MD, Professor of Pediatrics, University of North Carolina, Chapel Hill
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BB9998 Protocol 14; NHLBI P50-HL084934
Record Dates: First submitted 2009-06-17; First posted 2009-06-19 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-08

CONDITIONS: Healthy; Cigarette Smoking
Keywords: Otherwise healthy current cigarette smokers; current cigarette smokers
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endotoxin (Experimental): Inhalation of 20K EU CCRE
  Interventions: Biological: 20K EU CCRE

INTERVENTIONS:
Biological: 20K EU CCRE — Inhalation of CCRE

SUMMARY:
The purpose of this Phase 1 research study is to identify a dose of inhaled endotoxin that is safe (does not cause prolonged cough, shortness of breath or other problems), but causes changes in sputum cell samples that the scientists can measure. The investigators are also interested in seeing if the exposure to the endotoxin decreases the body's natural ability to clear mucus from the lungs.

DETAILED DESCRIPTION:
The purpose of this study is to determine the range of neutrophil response (influx of PMNs to the airways as determined in sputum) after inhalation of CCRE (20,000 EU), shown in previous studies of healthy, nonsmoking volunteers as well as in a limited number of otherwise healthy smokers to be well tolerated. This dose induces measurable increases in neutrophil content of induced sputum that can be employed to screen large populations for susceptibility to the inflammatory effect of inhaled endotoxin. Limitations of the understanding of actions of inflammatory stimuli on airway function are likely due to the fact that functional assessments of dynamic airway response /in vivo/ have generally been limited to those based on spirometry and examination of airway samples for assessment of cells and mediator content. Slowing of mucociliary clearance (MCC), a key component of airway defense, can be induced by inflammation and almost certainly contribute to mucus plugging and decreased clearance of inhaled irritants. Measures of mucociliary clearance (MCC), by inhalation of radiolabeled particles to label airway surface liquid, suggest that clearance of secretions is impaired to a mild degree in smokers and more severely in patients hospitalized for acute exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* Must be current cigarette smokers
* Must be otherwise healthy
* Must be good sputum producers

Exclusion Criteria:

* Any acute illness any chronic illness which would impact results

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Increase in sputum neutrophils | 6 hours

SECONDARY OUTCOMES:
Mucociliary clearance rates | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: David Peden, Principal Investigator — University of NC Chapel Hill Hospitals
Locations (1):
- UNC Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: Related Info — http://www.med.unc.edu/cemalb